CLINICAL TRIAL: NCT00236093
Title: A 4-week, Open-Label Extension Study of ACTIQ (Oral Transmucosal Fentanyl Citrate [OTFC]) Treatment for Opioid-Tolerant Children and Adolescents With Breakthrough Pain
Brief Title: Extension Study of ACTIQ Treatment for Children and Adolescents With Breakthrough Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C8278/2022/BP/US-CA
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Cancer; Sickle Cell Anemia; Severe Burns
Keywords: Sickle Cell
MeSH Terms: conditions — Pain; Neoplasms; Anemia, Sickle Cell; Burns | interventions — Fentanyl

INTERVENTIONS:
Drug: ACTIQ (Oral Transmucosal Fentanyl Citrate [OTFC])

SUMMARY:
The objective of the study is to monitor the safety (adverse event data) of longer-term use of ACTIQ (Oral Transmucosal Fentanyl Citrate [OTFC]) treatment in children with pain associated with cancer, sickle cell disease, or severe burns and breakthrough pain (BTP) who are receiving around the clock (ATC) opioid therapy.

ELIGIBILITY:
Inclusion Criteria:

Children are included in the study if all of the following criteria are met:

* The patient completed participation in ACTIQ double blind study in compliance with the protocol
* Written informed consent of the parent or legal guardian and patient assent, when appropriate, is obtained (lack of assent cannot be overturned)
* The child is aged 3 to under 16 years (at the time of enrollment into the ACTIQ double blind study) and continues to weight at least 15kg
* The child must continue using ATC opioid therapy for pain associated with cancer, sickle cell disease, or severe burns and be opioid-tolerant. Opioid tolerant patients are defined as patients who have taken at least 1 mg/kg/day or 40mg/day or more of oral morphine (or an equianalgesic dosage of another opioid) or at least 25 mcg/hour of transdermal fentanyl for at least 7 days. (ATC opioid therapy may be administered as patient controlled analgesia [PCA]).
* The child must be experiencing episodes of BTP (defined as transient flares of pain that require a bolus of medication as treatment) as follows:

  * Patients with cancer must be experiencing an average of at least 1 BTP episode a day
  * Patients with non-cancer related pain must be experiencing an average of 2 BTP episodes a day
* Girls who are postmenarch or sexually active must have a negative urine pregnancy test before entry into the study, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implanted, or injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence
* The child, in the opinion of the investigator, is able to administer ACTIQ treatment effectively (ie, adequately moving the unit around the mouth and sucking not biting the unit)
* The child may be an inpatient or outpatient

Exclusion Criteria:

Children are excluded from participating in this study if 1 or more of the following criteria are met:

* The child has pain uncontrolled by therapy, as determined by the investigator, that could adversely impact the safety of the patient or could be compromised by treatment with ACTIQ.
* The child has known or suspected hypersensitivities/allergies or other contraindications to any ACTIQ component
* The child has received monoamine oxidase inhibitors (MAOIs) within 14 days of the first dose of study drug administration
* The child has moderate to severe oral mucositis
* The child has a neuromuscular disease, significant renal impairment, or significant hepatic impairment as determined by the investigator
* The child has any other medical condition or is receiving concomitant medication/therapy that would, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise data collection
* The child is receiving any experimental drug/therapy. NOTE: Children may not be participating concurrently in another study when the other study requires experimental drug therapy.
* The child is receiving any other treatment that, in the opinion of the investigator, could interfere with the pain response
* A female patient of childbearing potential, is pregnant, or is lactating (any girl becoming pregnant during the study will be withdrawn from the study)
* The child has, in the opinion of the investigator, a development delay that would interfere with the use of ACTIQ therapy

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2006-10; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The objective of the study is to monitor the safety (adverse event data) of longer-term use of ACTIQ treatment in children with pain and BTP who are receiving ATC opioid therapy.

CONTACTS AND LOCATIONS:
Overall Officials: John Messina, Study Director — Cephalon
Locations (28):
- United States (26):
  - Children's Hospital of Arkansas, Little Rock, Arkansas
  - Childrens Hospital of Orange, Orange, California
  - Lucille Packard Childresns Hospital, Palo Alto, California
  - Connecticut Childrens Medical, Hartford, Connecticut
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Nemours Childrens Clinc, Jacksonville, Florida
  - St. Joseph's Childrens Hopsital, Tampa, Florida
  - Kapi'olani Medical Center, Honolulu, Hawaii
  - University Hospitals of Iowa, Iowa City, Iowa
  - David Center for Childrens Pain and Palliative Care, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Scottish Rite Children's Medical Center, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Tod Childrens Hospital, Youngstown, Ohio
  - Milton S Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Cancer and Blood Disorders Center, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - Sacred Heart Medical Center, Spokane, Washington
  - West Virginia Univeristy, Morgantown, West Virginia
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Iwk Health Center, Halifax, Nova Scotia, Canada
- San Jorge Childrens Medical, San Juan, Puerto Rico